CLINICAL TRIAL: NCT02666638
Title: Technical Development of up to 7T Magnetic Field Strength
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 14-01932
Record Dates: First submitted 2016-01-21; First posted 2016-01-28 (Estimated); Last update posted 2022-04-01 (Actual); Status verified 2022-03

CONDITIONS: Healthy
Keywords: Magnetic Resonance Imaging (MRI)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Volunteers (Active Comparator): MRI on up to a 7T scanner without contrast.
  Interventions: Other: Control Volunteers
- Clinical Patients (Experimental): MRI on up to a 7T scanner without contrast.+ 10 minutes of research development imaging added onto their clinical MRI scans.
  Interventions: Other: Clinical Volunteers

INTERVENTIONS:
Other: Control Volunteers — MRI on up to a 7T scanner without contrast.
  Arms: Control Volunteers
Other: Clinical Volunteers — One-hour MRI on up to a 7T scanner without contrast + 10 minutes of research development imaging using radio frequency (RF) coils
  Arms: Clinical Patients

SUMMARY:
The objective of this study is to determine whether these new image acquisition strategies and techniques using of up to 7T can produce meaningful structural and physiological information that can serve to improve our understanding of various disease processes in the clinical setting. 200 Control volunteers will be scanned for approximately one hour, without contrast, on up to 7T MRI scanner. 200 Study Participants will be scanned using newly developed imaging software or hardware that conforms to applicable FDA standards and recommendations. The data (images) for the Control and Experimental Group will be de-identified by the scan technologist and downloaded to a workstation within the Radiology Department for offline processing. These images will be reviewed by a trained Radiologist after the subject has departed.

ELIGIBILITY:
Inclusion Criteria:

* Healthy control volunteers, male and female, ages 18 and older (no history of chronic illness, concussion, malignancies, etc.)

Exclusion Criteria:

* Contraindications with MRI (e.g. pacemakers or ferromagnetic material near vital structures, etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2015-09-18 (Actual); Primary Completion 2022-03-24 (Actual); Study Completion 2022-03-24 (Actual)

PRIMARY OUTCOMES:
Change in signal to noise ratio using statistical analysis | 25 minutes
Change in spatial resolution using statistical analysis | 25 minutes
Change in Temporal Resolution using statistical analysis | 25 minutes
Change in Image Contrast using statistical analysis | 25 Minutes
Change in image homogeneity using statistical analysis | 25 minutes
Change in artifact reduction using statistical analysis | 25 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Yongxian Qian, MD, Principal Investigator — New York University Medical School
Locations (1):
- New York University School of Medicine, New York, New York, United States